CLINICAL TRIAL: NCT06832189
Title: Everolimus and Epoetin for Sustained Liver Transplant Tolerance (EVEREST)(ITN101ST)
Brief Title: EVR and EPO for Liver Transplant Tolerance
Acronym: EVEREST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN101ST
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant
Keywords: Everolimus; Liver Transplant; Epoetin alfa; Tacrolimus
MeSH Terms: interventions — Everolimus; Epoetin Alfa; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): Adult liver transplant recipients on a TAC-based IS regimen will transition from Tacrolimus (TAC) to Everolimus (EVR), receive five doses of epoetin alfa (EPO) and concurrently initiate phased withdrawal from EVR. Target accrual for the study is 20 subjects who receive any dose of EPO, and up to 20 donors.
  Interventions: Drug: Everolimus; Drug: Epoetin alfa

INTERVENTIONS:
Drug: Everolimus — The starting dose of EVR will be based on the maintenance TAC dose of the subject at study entry:
  1. EVR 1 mg PO BID if TAC dose is <=2 mg BID
  2. EVR 2 mg PO BID if TAC dose is 2.5-7 mg BID
  3. EVR 3 mg PO BID if TAC dose is >7 mg BID
  The dosage will be adjusted as needed to achieve and maintain EVR trough concentration of 5-8 ng/mL.
Drug: Epoetin alfa — The dose used in this study is 10,000 units SC every 8 weeks (at study weeks 16, 24, 32, 40 and 48) for five doses
  Other Names: EPO; Erythropoietin; Procrit

SUMMARY:
This is an open label, single-arm, multicenter phase 1b study of stable adult liver transplant recipients on a tacrolimus (TAC)-based immunosuppression (IS) regimen who will transition from TAC to Everolimus (EVR), receive five doses of EPO and concurrently initiate phased withdrawal from EVR.

The primary objective is to test the safety of administering Everolimus (EVR) and epoetin alfa (EPO) to induce operational tolerance in stable adult liver transplant recipients

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and provide informed consent
2. 1-10 years post-liver transplant
3. Tacrolimus-containing maintenance immunosuppression (IS) regimen without corticosteroid. Mycophenolate mofetil (MMF) dose must be <=2000 mg daily or mycophenolic acid (MPA) dose<=1440 mg daily (if on MMF or MPA). Tacrolimus level must be <8 ng/ml on the 2 most recent laboratory results within 3 months.
4. Gamma glutamyl transferase (GGT) and alanine transaminase (ALT) <= upper limit of normal (ULN)
5. Estimated glomerular filtration rate (GFR) >=40 mL/min/1.73 m^2 using the CKD-EPI 2021 equation
6. Female subjects of reproductive potential must have a negative pregnancy test upon study entry
7. Female subjects with reproductive potential, must agree to use Food and Drug Administration (FDA)-approved methods of birth control for the duration of the study
8. Subjects must have current vaccinations or documented immunity as per the Division of Allergy, Immunology, and Transplantation (DAIT) vaccine guidance for subjects in transplant trials
9. Negative result of most recent tuberculosis (TB) testing or appropriately completed latent tuberculosis infection (LTBI) therapy. Testing should be conducted using either a purified protein derivative (PPD) or interferon-gamma release assay (i.e., QuantiFERON-TB, T-SPOT.TB). Results from tests performed within 12 months prior to study entry are acceptable in the absence of any intervening exposure to TB. Subjects with a positive test for LTBI must complete appropriate therapy for LTBI. LTBI treatment regimens should be among those endorsed by the Centers for Disease Control and Prevention (CDC)
10. Negative FDA-approved test for human immunodeficiency virus (HIV) diagnosis at screening or as documented in medical record, up to 12 months prior to screening)
11. Negative hepatitis C antibody test at screening or as documented in medical record, up to 12 months prior to screening, in subjects without a history of hepatitis C. If there is a history of treated hepatitis C, then documentation of two consecutive negative hepatitis C virus (HCV) quantitative RNA polymerase chain reaction (PCR) tests separated by at least 3 months is required. Untreated subjects with positive HCV antibody and a single negative quantitative HCV RNA are eligible. Historical negative HCV RNA results are acceptable in the above two cases with positive HCV antibody
12. Negative hepatitis B surface antigen and negative hepatitis B core antibody in subjects without a history of hepatitis B virus (HBV) infection, up to 12 months prior to screening. Those with known hepatitis B infection or positive hepatitis B surface antigen or positive hepatitis B core antibody must be on antiviral therapy and have negative HBV DNA quantitative PCR at screening

Exclusion Criteria:

1. Inability of a subject to comply with study protocol
2. Any medical condition requiring chronic systemic corticosteroid, e.g., severe reactive airways disease. Use of inhaled steroids is not an exclusion
3. Autoimmune cause of liver disease (including autoimmune hepatitis (AIH), primary sclerosing cholangitis, primary biliary cirrhosis)
4. Diagnosis of rejection within 52 weeks prior to screening
5. Donor human leukocyte antigen (HLA) typing unavailable or inadequate for assigning donor-specific antibody (DSA)
6. Need for uninterrupted anticoagulation
7. Known active current or history of invasive fungal infection, or mycobacterial infection within 1 year prior to screening
8. Human immunodeficiency virus (HIV)-positive
9. Serious uncontrolled concomitant major organ disease
10. Recipient of non-liver solid organ or bone marrow transplant
11. Any infection requiring hospitalization and IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks
12. Malignancy within the last 5 years except treated basal and squamous cell cancer of the skin or treated in situ cervical cancer. History of hepatocellular carcinoma in the explanted liver is acceptable provided that

    1. the last alpha fetoprotein obtained within 3 months prior to liver transplantation was < 400 microg/L, and
    2. the recipients' explanted liver did not have evidence of increased risk of recurrent cancer, i.e., explant was within the Milan criteria, with no vascular invasion, and with no cholangiocarcinoma morphology
13. Neutropenia (absolute neutrophil count or ANC <1000 microliter) within 4 weeks prior to study enrollment
14. History of hypersensitivity to Epoetin (EPO) or mammalian Target of Rapamycin inhibitor (mTOR-I)
15. History of angioedema
16. History of hereditary disorders of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption. History of lactose intolerance is not an exclusion
17. History of genetic disorders predisposing to thrombosis including but not limited to Factor V Leiden mutation, prothrombin 20210, protein C deficiency, protein S deficiency, antithrombin III deficiency
18. History of venous or arterial thrombosis or thromboembolism, acute MI, or thrombotic stroke
19. History of Budd Chiari syndrome
20. Hemoglobin > 13.5 g/dl
21. Plasma fibrinogen or D-dimer level > ULN
22. Planned major surgery within the next 12 months
23. Uncontrolled severe hypertension
24. Uncontrolled clinically significant cardiac arrhythmia
25. Proteinuria with urine protein/creatinine >0.5 g/g
26. Severe hyperlipidemia with total cholesterol >350 mg/dl or triglycerides >1000 mg/dl
27. Current alcohol, drug, or chemical dependency
28. Currently pregnant or nursing
29. Current treatment with an estrogen-containing oral contraceptive, or systemic estrogen replacement therapy
30. Treatment with an immunomodulatory biological drug within 12 weeks of study entry
31. Immunization with live vaccine within 2 weeks of study baseline visit
32. Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational drug, whichever is longer) of screening
33. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the subject's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects free of opportunistic infection attributed to the investigational study regimen | At 52 weeks post-immunosuppression withdrawal (ISW)
  The primary analysis will be performed using the Intention-to-Treat (ITT) and Per-Protocol (PP) analysis populations, and the proportion will be summarized with a point estimate and a two-sided, 95% confidence interval (CI) calculated using the Clopper-Pearson (exact) method
The proportion of subjects free of malignancy attributed to the investigational study regimen | At 52 weeks post-immunosuppression withdrawal (ISW)
  The primary analysis will be performed using the Intention-to-Treat (ITT) and Per-Protocol (PP) analysis populations, and the proportion will be summarized with a point estimate and a two-sided, 95% confidence interval (CI) calculated using the Clopper-Pearson (exact) method
The proportion of subjects free of serious adverse events (SAEs) attributed to the investigational study regimen | At 52 weeks post-immunosuppression withdrawal (ISW)
  The primary analysis will be performed using the Intention-to-Treat (ITT) and Per-Protocol (PP) analysis populations, and the proportion will be summarized with a point estimate and a two-sided, 95% confidence interval (CI) calculated using the Clopper-Pearson (exact) method

SECONDARY OUTCOMES:
Incidence of acute rejection | From baseline to 156 weeks post-ISW completion
  All secondary endpoints (except for the change in eGFR) consider incidences or proportions, and therefore will follow the same analysis approach as the primary safety endpoint. Analysis will be performed using the Intention-to-Treat (ITT) and Per-Protocol (PP) analysis populations
  The proportion will be summarized with a point estimate and a two-sided, 95% confidence interval (CI) calculated using the Clopper-Pearson (exact) method.
Severity of acute rejection | From baseline to 156 weeks post-ISW completion
Timing of acute rejection | From baseline to 156 weeks post-ISW completion
Incidence of chronic rejection | From baseline to 156 weeks post-ISW completion
Severity of chronic rejection | From baseline to 156 weeks post-ISW completion
Timing of chronic rejection | From baseline to 156 weeks post-ISW completion
Incidence of de novo class II donor specific antibody (DSA) | From baseline to 156 weeks post-ISW completion
Incidence of graft loss | From baseline to 156 weeks post-ISW completion
Incidence of all-cause mortality | From baseline to 156 weeks post-ISW completion
Incidence of study-related Serious Adverse Event (SAE)s | From baseline to 156 weeks post-ISW completion
Incidence of opportunistic infections | From baseline to 156 weeks post-ISW completion
Incidence of malignancy | From baseline to 156 weeks post-ISW completion
Incidence of Everolimus (EVR) discontinuation due to Adverse Events (AEs) | From baseline to 156 weeks post-ISW completion
Incidence of polycythemia in the study | From baseline to 156 weeks post-ISW completion
Incidence of thromboembolism in the study | From baseline to 156 weeks post-ISW completion
Proportion of subjects with operational tolerance as defined by no rejection | At 52 weeks after completion of immunosuppression withdrawal (ISW)
  (clinical or biopsy-proven) since enrollment in the study and a liver biopsy demonstrating histologic stability and absence of rejection per the criteria delineated by the Banff Working Group on Liver Allograft Pathology [1], as assessed by the central pathology laboratory.
Change in estimated glomerular filtration rate (eGFR) | From baseline to 156 weeks after completion or failure of ISW
  Change in eGFR will be summarized using descriptive statistics (i.e., number of participants (n), mean, standard deviation (SD), median, first quartile (Q1), third quartile(Q3), minimum and maximum) at baseline, follow-up and for the change score. Follow-up scores will not be imputed. The ITT and PP analysis populations will be used.
Proportion of subjects with operational tolerance | At 156 weeks after completion of immunosuppression withdrawal (ISW)
Proportion of subjects who are clinically stable off immunosuppression (IS) | At 52 weeks after completion of immunosuppression withdrawal (ISW)
Proportion of subjects who are clinically stable off immunosuppression (IS) | At 156 weeks after completion of immunosuppression withdrawal (ISW)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Feng, MD, PhD, Study Chair — University of California, San Francisco; Paolo Cravedi, M.D., Ph.D., Study Chair — Icahn School of Medicine at Mount Sinai: Transplantation
Locations (3):
- United States (3):
  - University of California San Francisco School of Medicine, San Francisco, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: http://www.immport.org/home

REFERENCES:
- See also: Immune Tolerance Network (ITN) — https://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait